CLINICAL TRIAL: NCT05876819
Title: Comparison of Quality of Care and Welfare Services for Disabled Middle Older Adults in Iran Lebanon A Cross Sectional Study in 2023
Brief Title: Quality of Care and Welfare Services for Disabled Middle Older Adults in Iran Lebanon
Acronym: ServQual
Status: Enrolling by invitation | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Abdolrahim Asadollahi, PhD, Head of Dept. of Gerontology, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.SCHEANUT.REC.1402.03
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life; Health Care Acceptability; Disabilities Mental
Keywords: Older People; Middle Aged; Disabled; ServQual Model; IRAN; LEBANON; Quality of Services; Health System; Instrumentation; Quality of Caring
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iranians: Disabled Middle and Older Adults
- Lebanese: Disabled Middle and Older Adults

SUMMARY:
The findings of this research will be a basis for improving the quality of care and welfare services for the disabled middle-aged and older people in Iran and Lebanon using the SERVQUAL model.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 of years and above.
* Being Disabled.
* Receiving Health Care Services out of 1 year ago.

Exclusion Criteria:

* Unwillingness to Participate in the Study
* Death and/or Migration

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Iranian & Lebanese disabled mid/older adults who are received health care services from the local authorities out of 1 years ago.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ServQual | 8 Months
  Quality of Services to the Clients upon SERVQUAL Model

CONTACTS AND LOCATIONS:
Locations (1):
- Welfare Services Affairs, Shiraz, Dars, Iran

IPD SHARING:
Plan to Share IPD: Yes
Results and Data
Supporting Information: SAP, Analytic Code
Time Frame: June 2023 to Jan. 2024
Access Criteria: Sending email to Dr. Asadollahi